CLINICAL TRIAL: NCT06578065
Title: Colorectal Anastomosis Outcomes Using the Novel Powered Circular Stapler Compared With Manual Circular Staplers. A Randomized Multicentre Controlled Trial.
Brief Title: Colorectal Anastomosis Outcomes Using the Novel Powered Circular Stapler Compared With Manual Circular Staplers.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPCS-01-22
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Anastomosis

STUDY DESIGN:
Intervention Model Description: A multicenter, randomized, open-label, controlled with parallel groups clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ECPS group (Experimental): Echelon Circular™ Powered Stapler
  Interventions: Device: Echelon Circular™ Powered Stapler
- MCS Group (Active Comparator): 2-row circular staplers manual
  Interventions: Device: 2-row circular staplers manual

INTERVENTIONS:
Device: Echelon Circular™ Powered Stapler — Echelon Circular™ Powered Stapler will be used in colorectal anastomosis.
  Arms: ECPS group
Device: 2-row circular staplers manual — 2-row circular staplers manual will be used in colorectal anastomosis.
  Arms: MCS Group

SUMMARY:
Patients whom meet all eligibility criteria will be assigned random 1:1 to one of the following arms:

* ECPS group: Echelon Circular™ Powered Stapler (n=270)
* MCS Group: manual circular staplers (n=270) Patients will be followed during 30 days in order to evaluate the primary endpoint.

DETAILED DESCRIPTION:
Anastomotic Leakage (AL) is the complication that most concerns colorectal surgeons. It leads to prolonged postoperative stay, increased costs, risk of reoperations and a permanent colostomy, together with an increase in morbidity and mortality.

The novel Echelon Circular™ Powered Stapler (ECPS) (Ethicon, Somerville, NJ, USA), introduces design changes that could decrease the rate of technical errors and improve clinical outcomes. The powered stapler decreases the force needed on firing the device, improving stability at the anastomotic site. Atraumatic Gripping Surface Technology reduces the compressive forces on tissues, and along with 3D Stapling Technology allows a better compression distribution throughout the anastomosis and a better hemostasis.

This is a multicenter, randomized, open-label, controlled with parallel groups clinical trial, with 8 participant sites in total (4 sites in Spain and 4 sites in France), to include an approximate sample size (n) of 570 patients who will undergo a colorectal anastomosis after Hartmann reversal, left colectomy, sigmoidectomy or anterior rectal resection, for benign or malignant pathology.

540 patients assigned randomly 1:1 to assess whether technical improvements of Echelon Circular™ Powered Stapler (ECPS) have an impact on left-sided colorectal Anastomotic Leakage (AL) rate compared to current manual circular staplers (MCS).

Anastomosis could be performed open, laparoscopically or with robotic assistance.

After surgery, patients will be followed during 30 days in order to evaluate the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Patient or its legal representative informed consent.
* Age ≥ 18 years.
* Patients who will undergo a colorectal anastomosis after left colectomy, sigmoidectomy or anterior rectal resection, for benign or malignant pathology (NOTE: Hartmann reversal cases also included).

Exclusion Criteria:

* Diverting stoma.
* Emergency surgery.
* American Society of Anaesthesiologists (ASA) score ≥ IV.
* Transanal total mesorectal excision approach.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Anastomotic leakage rates differences between both groups at 30 postoperative days | Through study completion, an average of 1 year
  To assess whether ECPS have an impact on left-sided colorectal AL rate compared to current manual circular staplers (MCS).

SECONDARY OUTCOMES:
Postoperative endoluminal bleeding rate differences between both groups. | Through study completion, an average of 1 year
  To assess whether ECPS improve haemostasis in the anastomotic line
Morbidity differences between groups according to the Clavien-Dindo classification. | Through study completion, an average of 1 year
  To evaluate whether ECPS have an impact in postoperative morbidity
Re-intervention rate differences between both groups | Through study completion, an average of 1 year
  To evaluate whether ECPS have an impact in re-interventions rate

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Consorci Corporació Sanitària Parc Taulí de Sabadell, Sabadell, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Clínico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No